CLINICAL TRIAL: NCT01347060
Title: Outcomes for Medicare Asthma Patients Taking Fluticasone Propionate/Salmeterol Xinafoate Combination Versus Inhaled Corticosteroids or Other Combination Therapy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112605
Record Dates: First submitted 2010-06-10; First posted 2011-05-04 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma; treatment; Advair and inhaled corticosteroids; Medicare; Outcomes; costs
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medicare-eligible subjects with asthma: Asthma subjects at least 65 years of age enrolled in a large Medicare managed care health plan.
  Interventions: Drug: fluticasone propionate/salmeterol xinafoate combination; Drug: inhaled corticosteroids

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol xinafoate combination — Fluticasone propionate/salmeterol xinafoate combination for asthma, all doses (100mcg/50mcg, 250 mcg/50mcg and 500 mcg/50mcg)
  Other Names: Advair (TM)
Drug: inhaled corticosteroids — Inhaled corticosteroids: beclomethasone dipropionte, mometasone, fluticasone propionate, budesonide, and flunisolide

SUMMARY:
The objective of this study is to compare healthcare utilization and costs in Medicare-eligible asthma patients (aged >65) who receive fluticasone propionate/salmeterol xinafoate combination or inhaled corticosteroids in a typical clinical practice using a retrospective observational cohort study design of large managed care database. Outcomes on interest include asthma related severe exacerbations defined as asthma related emergency department visits, hospitalizations or combined emergency department/hospitalization. Other outcomes of interest include use of albuterol, oral corticosteroids and overall asthma related costs. Outcomes of interest will be compared between the two treatment cohorts (fluticasone propionate/salmeterol xinafoate combination or inhaled corticosteroids). Dichotomous outcomes (emergency visits, hospitalizations etc) will be compared using Cox regression hazards analysis assessing time to first event for each asthma related endpoint adjusting for differences in baseline demographics such as age, gender, previous asthma medication use, co morbidities, costs, and plan demographics. Total asthma related costs will also be compared using generalized linear models adjusting for baseline differences.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with asthma as determined by ICD-9 codes and asthma drug use
* at least 65 years of age
* prescription for an inhaled corticosteroid

Exclusion Criteria:

* a diagnosis of chronic obstructive pulmonary disease or
* a prescription for a chronic obstructive pulmonary disease treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Medicare-eligible subjects age 65 years and older with a diagnosis of asthma being treated with an inhaled corticosteroid
Sampling Method: Non-Probability Sample
Enrollment: 17448 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Fluticasone Propionate and Salmeterol: Participants aged 65-79 years with 15-24 months of continuous enrollment (12 months pre-index and 3-12 months post-index), with asthma diagnosis, and who received (index) Fluticasone Propionate and Salmeterol 100 micrograms (mcg)/50 mcg, 250 mcg/50 mcg, and 500 mcg/50 mcg
- Inhaled Corticosteroids: Participants aged 65-79 years with 15-24 months of continuous enrollment (12 months pre-index and 3-12 months post-index), with asthma diagnosis, and who received (index) Inhaled Corticosteroids (beclomethasone dipropionate, fluticasone propionate, mometasone furoate, triamcinolone, flunisolide, budesoninde). Due to the retrospective nature of this analysis, doses received and frequency of dosing are not known.
Period: Overall Study
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids
Started | 9868 | 7580
Completed | 9868 | 7580
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids | Total
Number analyzed (Participants) | 9868 | 7580 | 17448
Age, Customized [Number; unit: Participants]
  65-69 years old | 4153 | 3064 | 7217
  70-74 years old | 2694 | 2669 | 5363
  75-79 years old | 3021 | 1847 | 4868
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6083 | 4800 | 10883
  Male | 3785 | 2780 | 6565
Number of participants with comorbid COPD at baseline [Number; unit: participants] — International Classification of Disease-9 (ICD-9) codes 491, 492, 496, 490-492.8, 493.00-493.91, 494, 495.0-505, 506.4
  participants | 9227 | 7153 | 16380

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Post-index Asthma-related Events Measured Using Medical and Pharmacy Claims
Description: Asthma-related events were defined as events with any primary ICD-9 code of 493.xx for hospitalizations, emergency department visits, and combined hospitalization/emergency department visits. The post-index period is defined as 3-12 months after either the first administration of fluticasone propionate and salmetrol or inhaled corticosteroids. Medical and pharmacy claims are recorded healthcare encounters in a large managed care administrative insurance database.
Time Frame: Up to 7 years from July 1, 2001 to June 30, 2008
Population: Participants contributing to the PharMetrics database (a large, multiplan insurance encounter database) who were identified in the study as having at least one pharmacy claim for fluticasone propionate/salmeterol or inhaled corticosteroids, had an ICD-9 code of 493.xx for asthma, and were at least 65 years of age within the time frame of the study.
Measure: Mean (Standard Deviation); unit: Asthma-related events
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids
Number analyzed (Participants) | 9868 | 7580
Asthma-related events
  Inpatient visits | 0.033 (0.21) | 0.046 (0.25)
  Emergency department visits | 0.022 (0.18) | 0.027 (0.20)
  Inpatient/emergency department visits | 0.05 (0.30) | 0.07 (0.35)
Statistical Analysis 1: Comparison: Fluticasone Propionate and Salmeterol vs Inhaled Corticosteroids; Test type: Superiority or Other; p = 0.0051, Regression, Cox — The P-value relates to differences in combined inpatient/emergency department; Adjusted for baseline differences; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.68 to 0.93]

2. Secondary Outcome: Mean Asthma-related Costs in the Post-index Period
Description: Asthma-related costs were calculated as pharmacy costs, medical costs, and total asthma (pharmacy plus medical) costs. Medical costs were made up of asthma-related visits, hospitalizations, emergency department visits, and medical office visits. Pharmacy costs were comprised of all asthma-related medications used during the follow-up period. Medical services were identified by place of service and PharMetrics-specific confinement codes. Prescriptions were counted by 30-day fills, with fills less than 30 days rounded up to indicate one fill.
Time Frame: Up to 7 years from July 1, 2001 to June 30, 2008
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids
Number analyzed (Participants) | 9868 | 7580
United States dollars
  Medical Services Costs | 381 (2859) | 462 (2859)
  Pharmacy Costs | 1128 (1077) | 939 (1125)
  Total Asthma Costs | 1509 (3832) | 1401 (3151)
Statistical Analysis 1: Comparison: Fluticasone Propionate and Salmeterol vs Inhaled Corticosteroids; Test type: Superiority or Other; p = 0.001, Regression, Linear — The P-value is on the adjusted difference in total asthma costs; Generalized Linear Model with a log-link and a gamma distribution adjusting for differences at baseline; Mean Difference (Net) = 883.23, 95% CI 2-sided [731.66 to 1041.69]

3. Secondary Outcome: Mean Number of Albuterol (Short-acting β-Agonists) Canisters Dispensed Per Pharmacy Claim Per Participant
Description: The number of albuterol canisters dispensed was used as a surrogate marker of asthma symptoms.
Time Frame: Up to 7 years from July 1, 2001 to June 30, 2008
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: albuterol canisters
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids
Number analyzed (Participants) | 9868 | 7580
albuterol canisters | 1.01 (2.26) | 1.5 (2.95)
Statistical Analysis 1: Comparison: Fluticasone Propionate and Salmeterol vs Inhaled Corticosteroids; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: This was a retrospective observational study using a large health insurance claims database. Serious adverse events and non-serious adverse events were not collected.
Arm/Group | Fluticasone Propionate and Salmeterol | Inhaled Corticosteroids
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.